CLINICAL TRIAL: NCT05656573
Title: Phase I Study of CART-PSMA Cells in Patients With Advanced Prostate Cancer
Brief Title: CART-PSMA Cells for Advanced Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nova Therapeutics LLC (Industry)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NT1921-H301-CART-PSMA
Record Dates: First submitted 2022-12-01; First posted 2022-12-19 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- autologous CART-PSMA cells (Experimental): Cohort 1： CART-PSMA cells 1-3x10^7/M^2(body surface area) on Day 0; Cohort 2： CART-PSMA cells 1-3x10^8/M^2(body surface area) on Day 0; Cohort 3： Lymphodepletion chemotherapy with fludarabine (30 mg/m2 body surface area) plus cyclophosphamide (300 mg/m2 body surface area) for 3 consecutive days during D-7 to D-3, followed by the infusion of CART-PSMA cells at 1-3x10^7/M^2(body surface area) on Day 0.
  Cohort 4： Lymphodepletion chemotherapy with fludarabine (30 mg/m2 body surface area) plus cyclophosphamide (300 mg/m2 body surface area) for 3 consecutive days during D-7 to D-3, followed by the infusion of CART-PSMA cells at 1-3x10^8/M^2(body surface area) on Day 0.
  Interventions: Drug: CART-PSMA cells

INTERVENTIONS:
Drug: CART-PSMA cells — This study consists of 2 parts:
  Part A (Dose Escalation): The investigators are looking the highest dose of the study intervention that can be administered safely without severe or unmanageable side effects in participants that advanced prostate cancer.
  Part B (Expansion Cohort): Participants will be treated at the respective dose (at or below the Maximum Tolerated Dose), as determined during Part A (Dose Escalation).
  Up to 4 dosing cohorts, with up to 3 subjects enrolled in each cohort, will be explored as follows:
  Cohort 1： CART-PSMA cells 1-3x10^7/M^2 (body surface area); Cohort 2： CART-PSMA cells 1-3x10^8/M^2 (body surface area); Cohort 3： Lymphodepletion chemotherapy + CART-PSMA cells 1-3x10^7/M^2 (body surface area); Cohort 4： Lymphodepletion chemotherapy + CART-PSMA cells 1-3x10^8/M^2 (body surface area).
  Other Names: No other names

SUMMARY:
This is a single center, open-label phase 1 study to assess the safety and feasibility of PSMA-specific CAR modified autologous T cells (CART-PSMA cells) in patients with advanced prostate cancer.

DETAILED DESCRIPTION:
Part A (Dose Escalation) + Part B (Expansion Cohort) total up to 20 patients enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. All participants must have the ability to understand and the willingness to sign a written informed consent.
2. Histologic confirmation of prostate cancer.
3. Tumor expressing PSMA as demonstrated by immunohistochemistry analysis or other methods.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2.
5. Under general air conditions, blood oxygen saturation >90%.
6. Adequate liver function, specifically alanine aminotransferase (ALT) < 3 times of upper limit of normal (ULN), aspartate transferase (AST)< 3 times of ULN, serum bilirubin and alkaline phosphatase < 2 times of ULN.
7. Adequate renal function, specifically serum creatinine < 2.0 mg/dl.
8. Adequate cardiac function, specifically left ventricular ejection fraction (LVEF)≥50%.
9. Hemoglobin concentration ≥80g/L.
10. The side effects brought by the latest treatment should be recovered, and the latest chemotherapy should be at least 7 days before; At least three t½ have passed since the latest immunotherapy.

Exclusion Criteria:

1. Patients with other malignant tumors or major diseases.
2. Patients who are already undergoing other clinical drug trials or other gene therapy or cell therapy.
3. Patients with uncontrolled active infection.
4. Patients with active hepatitis B or hepatitis C infection.
5. Patients with human immunodeficiency virus (HIV) infection.
6. Patients who are being treated with immunosuppressive agents or systemic steroids (other than inhalation therapy).
7. Patients with various types of serious heart disease or a history of severe cerebrovascular disease.
8. Patients with congenital immune deficiency diseases or bone marrow deficiency diseases.
9. Patients with active autoimmune disease, including connective tissue disease, uveitis, inflammatory bowel disease, or multiple sclerosis; or a history of severe (as judged by the physician-investigator) autoimmune disease requiring prolonged immunosuppressive therapy.
10. Patients with active medical condition that, in the opinion of the physician-investigator, would substantially increase the risk of uncontrollable CRS (cytokine release syndrome) or CAR Neurotoxicity.

Ages: 35 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of study related adverse events, laboratory toxicities and clinical events that are possibly, likely, or definitely related to study participation. | Up to 15 years
  Assessing the type, frequency, severity, and duration of adverse events as a result of CART-PSMA cell infusion via physical, laboratory and imaging examination.

SECONDARY OUTCOMES:
The persistence, accumulation, and migration of CART-PSMA cells. | Up to 2 years
  Assessing the trafficking of CART-PSMA cells in the peripheral blood by quantifying the mRNA of CAR gene at the time of each infusion as well as at each time of follow-up blood collection. Peripheral blood will be collected prior to the initial infusion and will be set as baseline.
Overall survival (OS) | Up to 15 years
  Estimating median OS from CART-PSMA cell infusion to the event date (death) or last contact date (censor date) by Kaplan Meier methods.
Progression-free survival (PFS) | Up to 15 years
  Estimating median PFS by survival without biochemical (PSA) or radiographic evidence of disease progression or relapse from CART-PSMA cell infusion to event date (progression/relapse or death); the censor date: off protocol therapy date (required disallowed treatment or withdrawal of consent for further therapy) or last contact date.
Patterns of change in PSA (prostate-specific antigen) | Up to 5 years
  Assessing PSA response by the percentage of change in PSA from baseline to the defined time-frame on therapy (or earlier if patients discontinue therapy prior to the time-frame) as well as the maximum decline in PSA that occurs at any point during CART-PSMA cell infusion.
Serum cytokine profile | Up to 2 years
  Assessing potential cytokine release syndrome (CRS) toxicity and CART cell effector function, sequential serum samples by analysis of Th1/Th2 cytokines (e.g., IL-2, IFNgamma, TNFalpha, IL-10, GMCSF, IL-6, MIP-1alpha) before and after CART-PSMA cell infusion.
Phenotypes and frequencies of immune cell subsets in the peripheral blood pre- and post-therapy | Up to 2 years
  Assessing phenotypes and frequencies of immune cell subsets in the peripheral blood, T cell subsets and phenotypes utilising groups of labelled antibodies.
Changes in circulating tumor cells in peripheral blood | Up to 2 years
  Assessing changes in levels of circulating tumor cells (CTC) to investigate if decreases in CTC levels correlate with response.
Circulating cell-free deoxyribonucleic acid (cfDNA) in peripheral blood | Up to 2 years
  Assessing changes in levels of cfDNA to investigate if decreases in cfDNA levels correlate with response.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Zhang, Study Director — Nova Therapeutics LLC
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No